CLINICAL TRIAL: NCT03536026
Title: Localization of Peripheral Pulmonary Lesions: A Pilot Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Was unable to enroll any participants
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201711034
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Peripheral Lung Lesions
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bronchoscopic evaluation and biopsy (Experimental): -Bronchoscopy will be performed by pulmonary and/or critical care fellows who have performed fewer than 10 bronchoscopies (inexperienced bronchoscopists) under direct supervision by an attending Interventional Pulmonologist. The inexperienced bronchoscopist will attempt to navigate to the targeted peripheral pulmonary lesion without virtual bronchoscopic navigation, using only standard axial CT images as a reference. The attending physician will directly observe, but will provide no guidance during this period, which will last no longer than 10 minutes. If the lesion is located and confirmed with radial probe endobronchial ultrasound prior to 10 minutes, biopsies will be performed as per routine clinical practice. If the 10 minute time period elapses prior to localization of the peripheral pulmonary lesion, virtual bronchoscopic navigation will be used.
  Interventions: Procedure: Conventional bronchoscopy; Device: VIDA Pulmonary Workstation 2; Procedure: Biopsy

INTERVENTIONS:
Procedure: Conventional bronchoscopy — -Standard of care
Device: VIDA Pulmonary Workstation 2 — -Virtual bronchoscopic navigation system
Procedure: Biopsy — -Standard of care

SUMMARY:
Despite technological advancements directed towards the diagnosis of peripheral pulmonary lesions, an optimal approach has yet to be designed. One significant barrier for the bronchoscopic biopsy of peripheral lesions is the ability to reliably locate peripheral lesions in an efficient manner. The majority of the published literature regarding peripheral lesion biopsy has used diagnostic yield as the primary endpoint. Based on this data, it is unclear if non-diagnostic procedures are due to the inability to locate peripheral lesions, or due to the inability to successfully biopsy lesions once located using currently available instruments. This study will evaluate the bronchoscopists' ability to locate peripheral pulmonary lesions by using a conventional chest computed tomography (CT) scan as a reference and a virtual bronchoscopic navigational system, if needed, for the localization of peripheral pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral lung lesions 1-5cm in size identified on chest CT with the intention to undergo bronchoscopic evaluation and biopsy. The decision to pursue biopsy will be made by the treating physician and agreed upon by the patient.
* Are at least 18 years old
* Are able to provide informed consent
* Have CT scans within 30 days suitable for use with the virtual bronchoscopic system

Exclusion Criteria:

* Patients who refuse to participate
* Are less than 18 years of age
* Are pregnant
* Are physically unable to tolerate flexible bronchoscopy or moderate sedation as determined by the bronchoscopist
* Are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Localization of peripheral pulmonary lesions as confirmed using radial probe endobronchial ultrasound | At the time of bronchoscopy (day 1)

SECONDARY OUTCOMES:
Rate of lesion localization using a conventional chest CT as a reference only | At the time of bronchoscopy (day 1)
Rate of lesion localization using virtual bronchoscopic navigation if needed (failed lesion localization using conventional chest CT only) | At the time of bronchoscopy (day 1)
Time to localization of peripheral pulmonary lesions | At the time of bronchoscopy (day 1)
Diagnostic yield of procedures | At the time of bronchoscopy (day 1)
  -Diagnostic yield based on final cytology and/or histopathology will be determined from the results of the bronchoscopy. A biopsy that results in a specific diagnosis, either malignant or benign, that adequately explains the clinical scenario as determined by the treating physician, will be considered truly positive.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu